CLINICAL TRIAL: NCT04923841
Title: Effectiveness of Bright Light Therapy, Myopic Defocus, Atropine and the Combinations for Controlling Myopic Eye Growth in Schoolchildren: A Randomized Control Trial
Brief Title: Myopia Control Using Bright Light Therapy, Myopic Defocus and Atropine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R5032-18
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Myopia
Keywords: Myopia control; Bright light; Myopic defocus; Atropine
MeSH Terms: conditions — Myopia | interventions — Ultraviolet Therapy; Atropine; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (No Intervention): Subjects in control will receive single vision spectacle lenses and a placebo desk lamp
- BLT monotherapy (Experimental): Subjects in BLT monotherapy group will receive a high intensity light box for bright light therapy and single vision spectacle lenses
  Interventions: Other: High intensity light box for bright light therapy and single vision spectacle lenses
- BLT and DIMS (Experimental): Subjects in BLT and DIMS group will receive a high intensity light box for bright light therapy and Defocus Incorporated Multiple Segments (DIMS) spectacle lenses
  Interventions: Other: High intensity light box for bright light therapy and Defocus Incorporated Multiple Segments (DIMS) spectacle lenses
- BLT and atropine (Experimental): Subjects in BLT and atropine group will receive a high intensity light box for bright light therapy, single vision spectacle lens, and atropine 0.01% eye drop (twice a day)
  Interventions: Other: High intensity light box for bright light therapy and atropine 0.01% eye drop and and single vision spectacle lenses
- Atropine monotherapy (Experimental): Subjects in atropine group will receive atropine 0.01% eye drop (twice a day) and single vision spectacle lenses
  Interventions: Other: Atropine 0.01% eye drop and and single vision spectacle lenses

INTERVENTIONS:
Other: High intensity light box for bright light therapy and single vision spectacle lenses — High intensity light box for bright light therapy and single vision spectacle lenses
  Arms: BLT monotherapy
Other: High intensity light box for bright light therapy and Defocus Incorporated Multiple Segments (DIMS) spectacle lenses — High intensity light box for bright light therapy and Defocus Incorporated Multiple Segments (DIMS) spectacle lenses
  Arms: BLT and DIMS
Other: High intensity light box for bright light therapy and atropine 0.01% eye drop and and single vision spectacle lenses — High intensity light box for bright light therapy and atropine 0.01% eye drop and and single vision spectacle lenses
  Arms: BLT and atropine
Other: Atropine 0.01% eye drop and and single vision spectacle lenses — Atropine 0.01% eye drop and and single vision spectacle lenses
  Arms: Atropine monotherapy

SUMMARY:
The purpose of the study is to investigate the effect of bright light therapy, myopic defocus, atropine and the combination in myopia control in schoolchildren.

DETAILED DESCRIPTION:
The present study is a multi-arm randomised clinical trial with a 24-month duration. Subjects will be healthy Hong Kong Chinese schoolchildren with low to moderate myopia. The aims are to determine the clinical effectiveness of bright light therapy on inhibiting myopia progression in schoolchildren, and to determine whether combination therapy using bright light therapy (BLT) and myopic defocus is more effective than monotherapy.

Study population Seven hundred and sixty Hong Kong Chinese children (152 in each) of A. Control group, B. BLT only group, C. BLT and Defocus Incorporated Multiple Segments (DIMS) group, D. BLT and atropine 0.01% group) and E. Atropine 0.01% group aged 7-12 years old will be recruited. They must not have had prior or current myopia control treatment, have no ocular or systemic diseases/abnormalities that affect visual function, refractive development or spectacle lens wear, and no previous intraocular or corneal surgery. They must not have allergy to atropine.

The eligible subjects will be randomly assigned into one of the four groups. Their cycloplegic refraction and axial length will be monitored every six months for 2 years. The changes in refractive errors and axial length between groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Myopia of at least -0.75D (spherical equivalent) in both eyes
* Age at enrolment: 7-12 year; Hong Kong Chinese
* Astigmatism and anisometropia: 1.50D or less
* Spectacle corrected monocular visual acuity (VA): 0.0 logMAR or better
* Parents' understanding and acceptance of random allocation of grouping and masking
* Able to wear the prescribed spectacle, put on eye drop and undergo light therapy daily.

Exclusion Criteria:

* Eye disease or binocular vision problems (e.g., strabismus, amblyopia, oculomotor nerve palsies, corneal disease, etc.)
* Previous intraocular or corneal surgery
* Systemic disease that may affect vision, vision development (e.g. endocrine, cardiac and respiratory diseases, diabetes, Down syndrome, etc.)
* Allergy to atropine
* Previous gas permeable, soft bifocal, or orthokeratology contact lens wear or bifocal/PAL/specific myopic control spectacle wear or use of atropine or pirenzepine (longer than 1 month of wear)
* Previous or current participation in myopia control studies

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 579 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Cycloplegic Refraction Change in spherical equivalent refraction (SER) | Baseline and 2 years
  Change in cycloplegic SER (in diopter) will be measured using an open field autorefractor

SECONDARY OUTCOMES:
Axial length | Baseline and 2 years
  Axial length (mm) will be measured after cycloplegia using a non-contact optical biometer

CONTACTS AND LOCATIONS:
Overall Officials: Chi Ho To, PhD, Principal Investigator — School of Optometry, The Hong Kong Polytechnic University
Locations (1):
- Centre for Myopia Research, The Hong Kong Polytechnic University and Department of Ophthalmology, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hon Y, Chun RKM, Cheung BKK, Lam DMK, Kong ACW, Ho LM, Lam WC, Lam TC, Lam CS, Lian J, Morgan IG, To CH, Leung CKS, Tse DY. Effectiveness of bright light therapy and combination with myopic defocus for controlling myopic eye growth in schoolchildren: study protocol for a randomised controlled trial (phase 1). BMJ Open Ophthalmol. 2025 May 19;10(1):e002044. doi: 10.1136/bmjophth-2024-002044. PMID 40389302